CLINICAL TRIAL: NCT06223633
Title: PK Papyrus Covered Coronary Stent System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 078.CAR.2019.D
Record Dates: First submitted 2020-11-04; First posted 2024-01-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-01

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PK Papyrus Covered Coronary Stent System (Experimental): PK Papyrus Covered Coronary Stent System has been approved for use in the treatment of free perforations, defined as free contrast extravasation into the pericardium, in native coronary vessels or saphenous vein bypass grafts greater than or equal to 2.75mm in diameter.
  Interventions: Device: PK Papyrus Covered Coronary Stent System

INTERVENTIONS:
Device: PK Papyrus Covered Coronary Stent System — PK Papyrus Covered Coronary Stent System has been approved for use in the treatment of free perforations, defined as free contrast extravasation into the pericardium, in native coronary vessels or saphenous vein bypass grafts greater than or equal to 2.75mm in diameter.

SUMMARY:
The PK Papyrus Covered Coronary Stent System is a coronary stent being used at Methodist Dallas Medical Center for patients with coronary perforations.

DETAILED DESCRIPTION:
The FDA has approved the PK Papyrus Covered Coronary Stent System for use in patients being treated for acute perforations of native coronary arteries and coronary bypass grafts in vessels ranging from 2.5 to 5.0 mm in diameter, under a Humanitarian Device Exemption (HDE #H170004). Methodist Dallas Medical Center will use this device for treating the above-described patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute perforations of native coronary arteries and coronary bypass grafts in vessels 2.5 to 5.0 mm in diameter

Exclusion Criteria:

* Patients in whom antiplatelet agents or anticoagulation therapy is contraindicated.
* Patients with a known allergy or hypersensitivity to amorphous silicon carbide or any other compound of the system (siloxane-based polyurethane, L-605 cobalt chromium alloy including tungsten and nickel).
* Lesions that cannot be reached or treated with the system.
* Lesions with threatened or abrupt closure during attempted pre-dilation prior to stent implantation.
* Risk of treatment-related occlusion of vital coronary artery side branches.
* Uncorrected bleeding disorders.
* Allergy to contrast media.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Determining the number of the unanticipated adverse events related to the use of PK Papyrus Coronary Stent Graft System | Up to 10 years
  Number of patients with PK Papyrus being treated for acute perforations of native coronary arteries and bypass grafts in vessels.
Number of patients with the device | 10 years
  number of patients with success coronary artery and bypass grafts

CONTACTS AND LOCATIONS:
Overall Officials: Luis Bowen, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States